CLINICAL TRIAL: NCT06415110
Title: A Prospective Analysis of the Efficacy of Allosync Expand and Autograft Bone Graft in Open Lumbar Spinal Fusion
Status: Enrolling by invitation | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: Allosync Expand
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Spondylolisthesis, Grade 1
MeSH Terms: conditions — Spondylolisthesis; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Allosync Expand: All enrolled patients will received Allosync Expand at 1-3 contiguous levels (L1-S1).
  Interventions: Device: Allosync Expand

INTERVENTIONS:
Device: Allosync Expand — Allosync Expand is used in lumbar posterolateral arthrodesis at 1-3 contiguous levels (L1-S1)
  Other Names: Acceell Family of Products (Accell DBM 100, Accell TBM, A2i, and Accell Connexus)

SUMMARY:
The purpose of this study is to assess the radiographic and clinical outcomes of spinal fusion following use of Allosync Expand and autograft bone graft.

DETAILED DESCRIPTION:
This is a single site, prospective study with patients selected as study subjects from the Investigator's standard patient population who fulfill the Inclusion/Exclusion Criteria and agree to participate in the study. The study surgery is standard of care, with patients identified as requiring surgery prior to enrollment. The study surgery is lumbar posterior fixation with supplemental posterolateral fusion at from 1 to 3 levels. One side of the posterolateral fusion will be Allosync Expand (utilizing the BMA Angel kit to hydrate) and the other side to autograft bone (control).

ELIGIBILITY:
Inclusion Criteria:

1. At least 22years of age at the time of consent
2. Subject must have a documented diagnosis of spondylolisthesis up to Grade I. and have confirmed back and/or radicular pain with associated spinal stenosis as documented by conditions such as:

   1. Instability as defined by >3mm translation or >5 degree angulation
   2. Osteophyte formation of facet joints or vertebral endplates
3. Subject presents with one or more of the following:

   1. Radiculopathy
   2. Sensory deficit
   3. Motor weakness
   4. Reflex changes
4. Subject requires lumbar posterolateral arthrodesis at 1-3 contiguous levels (L1-S1).
5. The number of levels decompressed must equal the number of levels fused.
6. Subject must have been unresponsive to conservative care for at least 3 months prior to fusion surgery.
7. Subject must be willing and able to sign an informed consent document.
8. Subject must be willing and able to return for all follow-up visits, agree to participate in postoperative clinical and radiographic evaluations and comply with the required study regimen.

Exclusion Criteria:

1. Subject has had prior lumbar spine fusion surgery at any level.
2. Subject has greater than grade 1 spondylolisthesis of the lumbar spine.
3. Subject is pregnant or nursing or planning to become pregnant during the two years (24 months) following arthrodesis
4. Subject has an active local or systemic infection.
5. Subject is a prisoner
6. Patient has any condition (including malignancy), that in the opinion of the Investigator, would prohibit the patient from complying with and/or completing the protocol

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A patient who meets all inclusion criteria and none exclusion criteria will be enrolled in the study. A patient is considered enrolled upon placement of the Allosync Expand during the surgical procedure. If the surgeon decides intra-operatively not to utilize Allosync Expand, the patient will be considered a screen failure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Lumbar fusion rate assessed via CT | 12 months post surgery
  Lumbar fusion rate assessed via CT at 12 months post surgery

SECONDARY OUTCOMES:
Clinical outcome via neck visual analog scale (VAS) | 12 months post surgery
  Standard of care patient reported neck visual analog scale (VAS) will be used to evaluate patient pain. On a scale of 0 to 10 with a score of 0 being no pain and a score of 10 being worst pain. A low score means a better clinical outcome. A high score means a worse clinical outcome.
Clinical outcome via Overall Quality of Life (EQ-5D) EuroQol Research Foundation | 12 months post surgery
  Standard of care patient reported Overall Quality of Life (EQ-5D) EuroQol Research Foundation will be used to evaluate patient quality of life. On a scale of 3 levels: no problems, some problems, and extreme problems. With a score of "no problems" being no interference in quality of life and a score of "extreme problems" being a high interference in quality of life. "No problems" responses means a better clinical outcome. "Extreme problems" responses mean a worse clinical outcome.
Clinical outcome via PROMIS short form - Physical Evaluation | 12 months post surgery
  Standard of care patient reported PROMIS short form - Physical Evaluation will be used to evaluate patient physical function. On a scale of 5 levels: without any difficulty, with a little difficulty, with some difficulty, with much difficulty, and unable to do. With a score of "without any difficulty" being no interference in physical function and a score of "unable to do" being high interference in physical function. "Without any difficulty" means a better clinical outcome. "Unable to do" means a worse clinical outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Orthopaedic Surgeons, Southfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No